CLINICAL TRIAL: NCT05508711
Title: Comparability of Transesophageal Echocardiography and Continuous Mini-invasive FloTrac/Vigileo System (© Edwards Lifesciences) for the Determination of Cardiac Output in Three Different Positions During General Anesthesia
Brief Title: Comparability of Transesophageal Echocardiography and FloTrac/Vigileo System Three Different Positions
Status: Completed | Type: Observational
Sponsor: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Lucelia Fernandes Ricciardi, Principal Investigator, Université Libre de Bruxelles
Other Study IDs: B4062021000220
Record Dates: First submitted 2022-08-15; First posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Cardiac Output
Keywords: Cardiac output monitoring; Mini-invasive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: 1. st cardiac output measurement (horizontal supine position): Transesophageal echocardiographic cardiac output measurements, data recorded and in the meantime the data of the FloTrac system (© Edwards Lifesciences) monitor recorded also.
  2. nd cardiac output measurement (Trendelenburg position): The operating table was then tilted in - 30 ° Trendelenburg (head-down) position. Echocardiographic measurements and FloTrac system (© Edwards Lifesciences) data were recorded.
  3. rd cardiac output measurement: The patients were positioned from Trendelenburg to reverse-Trendelenburg, the above-described data were recorded again.
  Interventions: Device: FloTrac/Vigileo system (© Edwards Lifesciences) (Edwards Lifesciences, Irvine, CA) device
- Group 2: 1. st cardiac output measurement (horizontal supine position): Transesophageal echocardiographic cardiac output measurements, data recorded and in the meantime the data of the FloTrac system (© Edwards Lifesciences) monitor recorded also.
  2. nd cardiac output measurement (reverse Trendelenburg position): The operating table was then tilted in + 30 ° reverse Trendelenburg (head-up) position. Echocardiographic measurements and FloTrac system (© Edwards Lifesciences) data were recorded.
  3. rd cardiac output measurement: The patients were positioned from reverse Trendelenburg to Trendelenburg, the above-described data were recorded again.
  Interventions: Device: FloTrac/Vigileo system (© Edwards Lifesciences) (Edwards Lifesciences, Irvine, CA) device

INTERVENTIONS:
Device: FloTrac/Vigileo system (© Edwards Lifesciences) (Edwards Lifesciences, Irvine, CA) device — Concomitant cardiac output measurement with transesophageal echocardiography and with the FloTrac/Vigileo system (© Edwards Lifesciences) (Edwards Lifesciences, Irvine, CA) device in 3 different positions (horizontal supine, Trendelenburg and reverse Trendelenburg position).

SUMMARY:
The use of cardiac output monitoring to guide intraoperative fluid management and inotropic drugs as part of a hemodynamic therapy algorithm reduce the complication rate in major abdominal surgery. The FloTrac/Vigileo system (© Edwards Lifesciences) (Edwards Lifesciences, Irvine, CA) device estimate cardiac output by using arterial pulse contour analysis. The accuracy of FloTrac/Vigileo have been proven in patients with normal cardiac index. Most of studies regarding FloTrac/Vigileo were performed in patients in horizontal supine position, which is not usually the reality in the operation theater during abdominal surgery. Therefore, the investigators realized this monocentric prospective clinical trial to study the accuracy and trending ability of the fourth generation FloTrac/Vigileo system cardiac output estimation in three different positions (horizontal supine, Trendelenburg and reverse Trendelenburg positions) in anesthetized patients undergoing elective major abdominal surgery. The reference method of cardiac output measurement used was the transesophageal echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective pancreatic, bladder or liver surgery requiring invasive monitoring and Trendelenburg position during the procedure

Exclusion Criteria:

* age under 18 years
* weight under 40 kg
* preoperative left ventricular ejection fraction (LVEF) less than 45%
* severe heart valve disease
* known intra-and/or extracardiac shunt
* pulmonary hypertension
* preoperative circulatory shock with need for hemodynamic inotropic support
* redo surgery
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients without heart disease or hemodynamic instability scheduled for elective pancreatic, bladder or liver surgery requiring invasive monitoring and Trendelenburg position during the procedure.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
To verify the FloTrac/Vigileo's ability to estimate cardiac output (L/min) in horizontal supine position. | Baseline
  To study the fourth generation FloTrac/Vigileo system accuracy to estimate cardiac output (L/min) in horizontal supine position in anesthetized patients undergoing elective major abdominal surgery. The reference method of cardiac output (L/min) measurement used was the transesophageal echocardiography. The two cardiac output measurement techniques were assessed using Bland-Altman method.
To verify the FloTrac/Vigileo's ability to estimate cardiac output (L/min) in Trendelenburg position. | Baseline
  To study the fourth generation FloTrac/Vigileo system accuracy to estimate cardiac output (L/min) in Trendelenburg position in anesthetized patients undergoing elective major abdominal surgery. The reference method of cardiac output (L/min) measurement used was the transesophageal echocardiography. The two cardiac output measurement techniques were assessed using Bland-Altman method.
To verify the FloTrac/Vigileo's ability to estimate cardiac output (L/min) in reverse Trendelenburg position. | Baseline
  To study the fourth generation FloTrac/Vigileo system accuracy to estimate cardiac output (L/min) in reverse Trendelenburg position in anesthetized patients undergoing elective major abdominal surgery. The reference method of cardiac output (L/min) measurement used was the transesophageal echocardiography. The two cardiac output measurement techniques were assessed using Bland-Altman method.

CONTACTS AND LOCATIONS:
Overall Officials: Lucélia FERNANDES RICCIARDI, M.D., Principal Investigator — Université Libre de Bruxelles
Locations (1):
- Université Libre de Bruxelles, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vender JS. Clinical utilization of pulmonary artery catheter monitoring. Int Anesthesiol Clin. 1993 Summer;31(3):57-85. doi: 10.1097/00004311-199331030-00006. PMID 8375911
- [Background] Mayer J, Boldt J, Wolf MW, Lang J, Suttner S. Cardiac output derived from arterial pressure waveform analysis in patients undergoing cardiac surgery: validity of a second generation device. Anesth Analg. 2008 Mar;106(3):867-72, table of contents. doi: 10.1213/ane.0b013e318161964d. PMID 18292432 (Retraction: PMID 21451067 Anesth Analg. 2011 May;112(5):1074)
- [Background] McLean AS, Huang SJ, Kot M, Rajamani A, Hoyling L. Comparison of cardiac output measurements in critically ill patients: FloTrac/Vigileo vs transthoracic Doppler echocardiography. Anaesth Intensive Care. 2011 Jul;39(4):590-8. doi: 10.1177/0310057X1103900409. PMID 21823375
- [Background] Suehiro K, Tanaka K, Mikawa M, Uchihara Y, Matsuyama T, Matsuura T, Funao T, Yamada T, Mori T, Nishikawa K. Improved Performance of the Fourth-Generation FloTrac/Vigileo System for Tracking Cardiac Output Changes. J Cardiothorac Vasc Anesth. 2015;29(3):656-62. doi: 10.1053/j.jvca.2014.07.022. Epub 2014 Nov 14. PMID 25440654
- [Background] Maeda T, Hamaguchi E, Kubo N, Shimokawa A, Kanazawa H, Ohnishi Y. The accuracy and trending ability of cardiac index measured by the fourth-generation FloTrac/Vigileo system and the Fick method in cardiac surgery patients. J Clin Monit Comput. 2019 Oct;33(5):767-776. doi: 10.1007/s10877-018-0217-1. Epub 2018 Nov 7. PMID 30406422
- [Result] Pearse RM, Harrison DA, MacDonald N, Gillies MA, Blunt M, Ackland G, Grocott MP, Ahern A, Griggs K, Scott R, Hinds C, Rowan K; OPTIMISE Study Group. Effect of a perioperative, cardiac output-guided hemodynamic therapy algorithm on outcomes following major gastrointestinal surgery: a randomized clinical trial and systematic review. JAMA. 2014 Jun 4;311(21):2181-90. doi: 10.1001/jama.2014.5305. PMID 24842135